CLINICAL TRIAL: NCT04653428
Title: German Registry for Transcatheter Tricuspid Valve Interventions
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other); Heart Center Leipzig - University Hospital (Other); Mainz University (Other); Universitätsklinikum Köln (Other); University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Jörg Hausleiter, Professor, LMU Klinikum
Other Study IDs: D-TRIK
Record Dates: First submitted 2020-11-17; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Insufficiency; Heart Valve
Keywords: Tricuspid regurgiation; Tricuspid valve insufficiency; Interventional treatment; Heart valve diseases
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

INTERVENTIONS:
Device: Interventional treatment of tricuspid regurgitation — Interventional treatment for tricuspid regurgitatin with CE-certified products, e.g. edge-to-edge repair

SUMMARY:
Multicentre observational study of patients with severe tricuspid regurgitation and interventional treatment.

DETAILED DESCRIPTION:
Severe tricuspid regurgitation occurs in around 1.5 % of men and 5.6 % of women and it is associated with significant morbidity and mortality. Current guidelines recommend cardiac surgery, especially in those patients who are undergoing left side valve surgery. Nevertheless many patients are not eligible for surgical tricuspid valve repair due to an high risk of mortality. Therefore interventional devices for treatment of tricuspid regurgitation have been established to offer these patients an alternative treatment option. The aim of this study is to analyse the success and saftey aspects of different interventional repair techniques for severe tricuspid regurgitation. Therefore in this prospectively designed observational study clinical, echocardiographic and laboratory parameters will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Interventional treatment of severe tricuspid regurgitation (isolated or in combination with another interventional treatment) with a CE certified product for tricuspid valve repair
* Informed consent corresponding to criteria of Good Clinical Practice and the decleration of Helsinki as well as to standards of the local ethic commission.

Exclusion Criteria:

* No agreement to participation
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe symptomatic tricuspid regurgitation, who are not eligible for cardiac surgery due to a high risk of mortality.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death and heart failure hospitalisation | 1 year
  All-cause death and heart failure hospitalisation 1 year after transcatheter tricuspid valve treatment (TTVT)

SECONDARY OUTCOMES:
All-cause death and heart failure hospitalisation (long-term) | up to 5 years
  Long-term all-cause death and heart failure hospitalisation after transcatheter tricuspid valve treatment (TTVT)
All-cause death and heart failure hospitalisation (short-term) | 30-90 days
  Short-term all-cause death and heart failure hospitalisation after transcatheter tricuspid valve treatment (TTVT)
Change of tricuspid regurgitation after transcatheter tricuspid valve treatment (TTVT) | up to 5 years
  Assessed by echocardiography, tricuspid regurgitation graded on a 4-grade scale.
Change of cardiopulmonal symptoms after transcatheter tricuspid valve treatment (TTVT) | up to 5 years
  Assessment for cardiopulmonal symptoms include edema scaling
Change of NYHA classification after transcatheter tricuspid valve treatment (TTVT) | up to 5 years
  NYHA classification I, II, III or IV
Change of 6-minute walking distance test after transcatheter tricuspid valve treatment (TTVT) | up to 5 years
  Assessed by standardized protocol testing 6-minute walking distance
Change of quality of life after transcatheter tricuspid valve treatment (TTVT) | up to 5 years
  Quality of life is assessed by standardized questionnaires including the Minnesota Living with Heart Failure Questionnaire
Change of NT-proBNP after transcatheter tricuspid valve treatment (TTVT) | up to 5 years
  N-terminal pro Brain Natriuretic Peptide (NT-proBNP) in pg/ml
Procedural success after transcatheter tricuspid valve treatment (TTVT) | At the day of discharge after transcatheter tricuspid valve treatment (TTVT)
  Procedural success is defined as a reduction of the tricuspid regurgitation to at least grade 2+ achieved by interventional treatment

OTHER OUTCOMES:
Safety outcome after transcatheter tricuspid valve treatment (TTVT) | At the day of discharge after transcatheter tricuspid valve treatment (TTVT)
  The saftety outcome contains all complications which occur between the interventional treatment of the tricuspid regurgitation and discharge from the hospital. Data collection includes: mortality with differentiation of cardiac death and non-cardiac death, unplanned cardiac surgery, re-intervention of tricuspid valve, pericardial tamponade, intervention of coronary arteries. Moreover major adverse events as defined by MVARC2 criteria are recorded at discharge from hospital: death with differentiation of cardiac death and non-cardiac death, peri-procedural or spontaneous myocardial infarction, stroke, transient ischemic attack, life-threatening, major or minor bleeding, acute kidney failure, complications of the vascular access.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Hausleiter, MD, Principal Investigator — Klinikum der LMU Muenchen
Locations (1):
- Klinikum der LMU Muenchen, Munich, Germany